CLINICAL TRIAL: NCT02851082
Title: Protected by Nature: Could Physical Activity Help to Counteract the Blood Haemophilia Disturbance? A Pilot Study.
Brief Title: Could Physical Activity Help to Counteract the Blood Haemophilia Disturbance? A Pilot Study.
Acronym: END-HEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15 7674 03
Record Dates: First submitted 2016-07-27; First posted 2016-08-01 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Hemophilia A
Keywords: Training Program; Endurance; Von Willebrand factor
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Haemophilia A patients (Experimental): Patients will perform endurance training program on 6 consecutive weeks
  Interventions: Other: Endurance training program

INTERVENTIONS:
Other: Endurance training program — Exercise intensity will be fixed to the corresponding powers for ventilatory thresholds, if applicable for pain tolerance. The endurance interval training workout is known to induce metabolic and physiological adaptations. For intermittent workout training protocol, recovery periods at moderate intensity between periods at high intensity help to sustain repeated high intensity periods of exercise. If pain disturbs exercise tolerance, power will be lowered as necessary.
  A set of 3 training sessions per week of 45 minutes each for 6 consecutive weeks will be proposed (one session every two days). This scheme is usually encouraged for patients suffering from chronic diseases.

SUMMARY:
Physical activity is lower in patients with haemophilia than in their healthy peers. Nevertheless, exercize is recommended for those patients and supported by evidence. Until 2013, scientific and medical evidence to encourage physical activity for patients with haemophilia were listed to increase their locomotor function, their metabolic status, their fitness level and their well-being. In 2013, an original publication by Groen et al. suggested that physical activity could also interact with the specific and biological disturbance of the disease.

We propose to consider that regular endurance exercize prescription should be encouraged in patients with haemophilia not only for a healthier lifestyle but also because it could positively alter the specific biological blood disturbance seen in haemophilia. Nevertheless, before planning a well powered intervention trial we need to determine the acceptability of regular exercize and the expected value of factor Factor VIII, von Willebrand factor and von Willebrand propeptide after an endurance training program.

ELIGIBILITY:
Inclusion Criteria:

* Mild (FVIII:1-5%) and moderate (FVIII:6-40%) haemophilia A patients,
* Living in the Midi-Pyrenees region,
* Between 18 and 45 years old,
* Exempt from any significant medical condition that could prevent them from being subjected to an endurance training program,
* Affiliated to a social security cover

Exclusion Criteria:

* Women
* Subjects declaring 2 or more spontaneous bleeding events and/or 4 or more induced bleeding events out of a traumatic circumstance 6 months prior to inclusion
* Absence of signed consent
* Patient protected by Justice

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Determine the acceptability of a 6-weeks endurance training program in patients with haemophilia A as assessed by specific clinical follow-up | During 6 weeks

SECONDARY OUTCOMES:
Variation of Factor VIII in response to acute exercise before and after the endurance training program as assessed by specific bioassay | Day 1 and after 6 weeks of training program
Variation of von Willebrand Factor in response to acute exercise before and after the endurance training program as assessed by specific bioassay | Day 1 and after 6 weeks of training program
Variation of von Willebrand propeptide in response to acute exercise before and after the endurance training program as assessed by specific bioassay | Day 1 and after 6 weeks of training program
Variation of maximal oxygen uptake in response to acute exercise before and after the endurance training program as assessed by specific endurance testing | Day 1 and after 6 weeks of training program
Variation of VO2max in response to acute exercise before and after the endurance training program as assessed by specific endurance testing | Day 1 and after 6 weeks of training program
Variation of quality of life of patients in response to acute exercise before and after the endurance training program as assessed by Haem-A-QoL questionnaire | Day 1 and after 6 weeks of training program
  The Haem-A-QoL questionnaire was specifically designed for adults with haemophilia

CONTACTS AND LOCATIONS:
Overall Officials: Fabien PILLARD, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided